CLINICAL TRIAL: NCT07153159
Title: A PHASE 1 MULTIPLE-DOSE, OPEN-LABEL PHARMACOKINETIC STUDY OF ETRASIMOD IN HEALTHY LACTATING WOMEN
Brief Title: A Study to Learn How the Study Medicine Called Etrasimod is Taken up Into Blood and Breastmilk of Healthy Breastfeeding Women
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: C5041053; 2025-520930-44-00 (Registry Identifier: CTIS (EU))
Expanded Access: NCT06025227 (Available)
Record Dates: First submitted 2025-08-05; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Healthy Participant
Keywords: Breast feeding women
MeSH Terms: interventions — etrasimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- healthy breast feeding volunteers (Experimental)
  Interventions: Drug: Etrasimod

INTERVENTIONS:
Drug: Etrasimod — Oral 2 milligrams tablet, once a day for 7 days

SUMMARY:
This study aims to figure out how much etrasimod, a medication, ends up in breast milk after taking it for several days. To do this, the researchers will work with at least 8 healthy women who are breastfeeding. These women will take a 2 mg dose of etrasimod every day for 7 days while staying at the testing site. During the study, they won't be allowed to breastfeed their babies to keep the babies safe. Instead, they need to have another plan for feeding their babies during this time. The study will look at how the medication is absorbed and how it moves through the body, checking things like the highest level in the blood and how long it takes to reach that level. The researchers will also see how much of the drug is in the breast milk compared to the blood and whether it's safe for the women to take. After the last dose, the women will stay at the site for at least another 24 hours before going home, and follow-up safety calls will be made about 14 and 28 to 35 days later. The whole process from start to finish will take about 10 weeks

ELIGIBILITY:
Inclusion

1. Healthy (as determined by medical evaluation including medical history, physical examination, laboratory tests, vital signs and 12-lead ECGs) lactating women who are actively breastfeeding or expressing breast milk, who are at least 12 weeks post partum and not currently pregnant (must have a negative pregnancy test), and must be 18 to 55 years of age, inclusive, at the time of signing the informed consent document (ICD).
2. Body mass index (BMI) of 16-35 kg/m2; and a total body weight >45 kg (99 lb).
3. Participants must be willing to temporarily discontinue breastfeeding their infants for a total of 21 days, ie, from the evening of the day before Day 1 through to 14 days after the last dose (approximately 8 AM the morning of Day 21). Participants must be willing to regularly pump breasts throughout the study and express breast milk according to a schedule designed to maintain lactation until the completion of breast milk collection

Exclusion

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary (such as moderate or severe chronic pulmonary disorders like asthma or chronic obstructive pulmonary disease [COPD]), gastrointestinal, cardiovascular, hepatic, neurological/psychiatric, anaphylactic, ophthalmologic disorders (such as macular edema, uveitis, retinopathy), or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
2. Participants with history or presence of second-degree or third-degree atrioventricular (AV) block, sick sinus syndrome, or sinoatrial block.
3. Resting HR <50 bpm at Screening or pre-randomization on Day 1. Measurement can be repeated up to 3 times to confirm the finding. Mean values will be used if repeated.
4. Recurrent symptomatic bradycardia or recurrent cardiogenic syncope
5. Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy).
6. Known immunodeficiency disorder, including positive serology for human immunodeficiency virus (HIV), or a first degree relative with a hereditary immunodeficiency, and history of organ transplant (except corneal transplant).
7. History or evidence of hepatitis B or hepatitis C viruses. Hepatitis B vaccination is allowed.89.
8. Participants with any of the acute or chronic infections or infection history

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female participants
Enrollment: 8 (Estimated)
Dates: Start 2025-08-07 (Actual); Primary Completion 2026-09-12 (Estimated); Study Completion 2026-10-12 (Estimated)

PRIMARY OUTCOMES:
Area under the etrasimod concentration-time curve in breast milk | Baseline (Day -1), Day 1, Day 7 and Day 8.
Maximum observed concentration of etrasimod in breast milk | Baseline (Day -1), Day 1, Day 7 and Day 8.
Amount of etrasimod excreted in breast milk | Baseline (Day -1), Day 1, Day 7 and Day 8.
Percent of etrasimod dose excreted in breast milk | Baseline (Day -1), Day 1, Day 7 and Day 8.
Breast milk clearance of etrasimod | Baseline through Day 8
  Baseline (Day -1), Day 1, Day 7 and Day 8.
Time to maximum observed concentration of etrasimod | Baseline (Day -1), Day 1, Day 7 and Day 8.

SECONDARY OUTCOMES:
Area under the etrasimod concentration-time curve in plasma | Day 1 hour 0, Day 7 hour 0, 1, 2, 4, 6, 8 and 12, Day 8 hour 24
Maximum observed concentration of etrasimod in plasma | Day 1 hour 0, Day 7 hour 0, 1, 2, 4, 6, 8 and 12, Day 8 hour 24
Time to maximum observed concentration of etrasimod in plasma | Day 1 hour 0, Day 7 hour 0, 1, 2, 4, 6, 8 and 12, Day 8 hour 24
Breast milk to plasma ratio for area under the concentration-time curve | Baseline (Day -1), Day 1, Day 7 and Day 8.
percentage of treatment emergent adverse events in participants | Baseline through Day 35
Number of Participants With Clinically Significant Change From Baseline in Laboratory Abnormalities | Baseline through Day 8
Number of Participants With Clinically Significant Change From Baseline in vital signs (blood pressure and heart rate) | Baseline through Day 8
Number of Participants With Clinically Significant Changes From Baseline in 12-Lead Electrocardiogram (ECG) Parameters | Baseline through Day 8
Body weight normalized infant dose in μg/kg/day | Baseline through Day 8
Body weight normalized maternal dose in μg/kg/day | Baseline through Day 8
Infant dose expressed as % of body weight normalized maternal dose | Baseline through Day 8

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - Brussels, Brussels, Bruxelles-capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5041053